CLINICAL TRIAL: NCT04467632
Title: Circadian & Homeostatic Synchronization Effect on Waking Mobility in Parkinson's Disease: a Feasibility Study
Brief Title: Circadian & Homeostatic Synchronization Effect on Waking Mobility in Parkinson's Disease
Acronym: Synch Fit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator left the hospital
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19_RIPH2-12
Record Dates: First submitted 2019-10-14; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Sleep benefit; circadian process; homeostatic process; circadian and homeostatic synchronization
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients affected with idiopathic Parkinson Disease (Experimental)
  Interventions: Other: Validation of the mobility assessment by IMU wearable sensors; Other: Testing in real-life conditions at patients' home in a small group of subjects

INTERVENTIONS:
Other: Validation of the mobility assessment by IMU wearable sensors — The validity of the mobility assessment by IMU wearable sensors will be verified in Work Package 3.
  It will be defined as the accuracy of the machine learning algorithm to predict patients' motor status compared to the motor status assessed at clinical examination by means of the MDS-UPDRS-III scale and the Fit test. Prediction by machine learning will be compared with the MDS-UPDRS-III total score and with the 3.14 item (global clinical impression of mobility) of the same scale.
  The patients will be asked to perform all the motor tasks of the MDS-UPDRS-III scale and the finger tapping test (Fit test) with both hands wearing the IMU system. A subset of minimal motor tasks allowing good prediction of the patient's motor status by the machine learning algorithm will then be selected for Work Package 4.
Other: Testing in real-life conditions at patients' home in a small group of subjects — Baseline Phase B1: Observation phase: 1-week wrist actigraphy and sleep diary to assess habitual activity/rest routines.
  B2: Nocturnal sleep consolidation phase: 2 weeks: timed light exposure, constant sleep/wake routine and sleep restriction of 1 hour/night (based on habitual activity).
Other: Testing in real-life conditions at patients' home in a small group of subjects — Intervention phase
  * Phase A (11 days): subjects will receive one hour of morning and afternoon light exposure twice a day:
    * Day #1: baseline assessment of outcome measures;
    * Days #2 to #6: bright light in the morning (active treatment) + dim light in the afternoon (placebo), to progressively advance circadian phase of 30' per day (phase advance of 2.5 hours obtained at day 6);
    * Days #7 to #11: dim light in the morning + bright light in the afternoon to revert the circadian phase to the baseline of 30' per day.
  * Washout: 6 days. No intervention during this phase, to stabilise the reverted circadian rhythm to baseline, for phase B to be held at the same conditions as phase A.
  * Phase B (11 days): similar as in phase A:
    * Day #1: similar as in phase A;
    * Days #2 to #6: reverted conditions compared to phase A.
    * Days #7 to #11: reverted conditions compared to phase A.

SUMMARY:
Sleep benefit (SB) consists of a spontaneous, transient and inconsistent improvement of the mobility occurring on morning awakening in approximately 40% of Parkinson's disease (PD) patients, before taking the first morning dose of dopaminergic drugs.

The SB could represent a pathway for the development of new therapeutic strategies for motor symptoms in PD.

Being a seemingly unpredictable phenomenon and a great variability daily, inter- and intra-subject, the SB study requires multiple and repeated assessments of mobility for several days. An experimental home setting would be optimal for this purpose in terms of cost-effectiveness and patient acceptability.

In addition, since the extent and nature of SB have not been well characterized so far, and the magnitude of its variability is unknown, a reliable assessment method, independent of observers and situation, the SB is a requirement of further research in this area.

A recently developed technique combining machine learning algorithms with wireless portable sensors (accelerometers and gyroscopes) and software applications could be particularly promising for characterizing the complexity and multiplicity of SBs in. With this technique, repeated and multiple assessments of mobility can be performed in the homes of patients without the constant presence of a researcher.

This approach offers several advantages in terms of cost-effectiveness, feasibility and acceptability of study protocols by patients. It also improves the ecological validity of subjective and objective estimates of mobility in these patients.

The investigators chose to conduct this preliminary study on patients with PD rather than on healthy subjects, because SB is a phenomenon that has been described so far only in this population. Investigators also consider that the feasibility of the study will depend mainly on the patients' ability to move and the context of their own illness.

SB is a phenomenon induced by sleep. The propensity and timing of sleep depend on the coordinated interaction of the duration of the previous awakening (homeostatic process) and a circadian signal (circadian process). In order to better understand SB, it is necessary to study the reciprocal influences of the circadian and homeostatic process.

Investigators have devised a new paradigm to "shift" the circadian process phase around the homeostatic process, maintained under constant conditions, in order to observe the effect of the synchronism or desynchronization of these two processes on the awakening mobility of patients with an MP. This experimental approach was approved by Professor Aleksandar Videnovic (Harvard University School of Medicine, USA), opinion leader on circadian rhythmicity in the MP and scientific collaborator of this study.

As a first step, the investigators plan to implement a technology-assisted home-based methodology, to validate it in PD patients and to verify the logistic feasibility of this method-assisted approach in a small group of patients, in order to to be able to apply this paradigm in larger scientific projects.

DETAILED DESCRIPTION:
Parkinson's disease is a common neurodegenerative disorder touching 1.5% of the general population over 60 year-old and featuring impaired mobility with high impact on daily living and quality of life of the patients and their caregivers. Fourty percent of the patients with Parkinson's disease (PD) report inconstant, prominent, spontaneous, transitory improvement in mobility occurring on morning awakening, before taking their first morning dose of dopaminergic medications. This apparently unpredictable, highly variable, sleep-related phenomenon has been named "Sleep Benefit" (SB) by the scientists.

SB is a promising track to follow to develop novel therapeutic strategies for motor symptoms in PD. An innovative approach could be to induce modifications of mobility by influencing sleep regulation in PD patients in experimental settings.

Sleep propensity and timing depend on the coordinated interaction of the duration of preceding wakefulness (homeostatic component) and on a circadian signal (circadian component). Reciprocal interactions between homeostatic and circadian processes preside to internal synchrony of many physiological processes. We hypothesize SB to depend on serendipitous optimal synchronization between circadian and homeostatic process on morning awakening. As SB shows high day-to-day, inter- and intra-subject variability, studying SB requires multiple, repeated assessment of mobility during several days. A home-based experimental setting would be optimal for this purpose in terms of cost-effectiveness and acceptability by the patients. Moreover, considering that the range and nature of SB has not been well characterized so far, and that the amplitude of its variability is unknown, a reliable, observer- and situation-independent, reproducible assessment method of SB is a pivotal requirement for further research in this area.

A recently developed technique associating machine-learning algorithms with wireless wearable sensors (accelerometers and gyroscopes) and software applications might be particularly promising to characterize the complexity and multiplicity of SB in PD. Thanks to this technique, repeated, multiple assessments of mobility can be performed at patients' home without the constant presence of an investigator.

The working hypothesis of this study is that motor performance in PD patients improves on morning awakening when optimal synchrony between circadian and homeostatic regulation of sleep occurs. As first step, we envision to set up a home-based and technology-assisted methodology and to verify its scientific, technological and logistic feasibility.

The study will involve four work packages, for each of which specific endpoints are defined:

WP1: Definition of the logistics, setting, practices of the study procedures for home assessment;

WP2: Technological setup of:

* IMU wearable sensors
* SleepFit software application development
* light therapy (included sham light therapy)
* home polysomnography
* chronobiological assessments (distal-proximal skin body temperature gradient; Dim Light Melatonin Onset (DLMO) from salivary specimens;

Two work packages (3 and 4) will require patients inclusion and interventions on patients:

WP3: Validation of mobility assessment by wearable sensors: accuracy of machine learning algorithm to predict patients' motor status based on the MDS-UPDRS-III total score and on the 3.14 item (global clinical impression of mobility);

WP4: Testing in real-life conditions at patients' home in a small group of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old;
* Patients affected with idiopathic PD, of both sexes;
* Hoehn and Yahr stage of 2 to 4 in the "on" state;
* Stable antiparkinsonian and/or psychotropic medications for at least 4 weeks prior to study screening;
* Reliable partner/caregiver to assist the patient during the study procedures;
* Affiliated person or beneficiary of a social security scheme;
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patients < 18 years old;
* Atypical parkinsonian syndromes;
* Dementia;
* Treatment with extended-release dopaminergic drugs (excluding extended release levodopa given no later than 6 hours before the habitual bedtime);
* Use of hypno-sedative drugs or stimulants;
* Use of antidepressants unless on a stable dose for at least 3 months;
* Travel through 2 time zones within 90 days prior to study screening;
* Visual abnormalities that may interfere with light therapy, such as significant cataracts, narrow angle glaucoma or blindness;
* Any other medical condition potentially interfering with the assessment of mobility (e.g. limb amputation, post-stroke paralysis, severe osteo-articular condition);
* Any condition limiting the capability of the subject to understand the task to be performed at home by the patient himself (e.g. aphasia, oligophrenia);
* Severely altered physical and/or psychological health which, according to, the investigator, could affect the participant's compliance of the study;
* Inadequate housing conditions to perform home assessments;
* Patients refusing to participate in the study;
* Patients under legal guardianship or curatorship, pregnant and breastfeeding women, women of child-bearing age, persons in emergency situations;
* Persons participating in another research including a period of exclusion still in course and at any case < 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Validation of the objective metrics of mobility | 12 months
  The validity of the mobility assessment by Inertial Measurement Unit (IMU) wearable sensors will be verified.
  It will be defined as the accuracy of the machine learning algorithm to predict patients' motor status compared to the motor status assessed at clinical examination by means of the MDSUPDRS- III scale and the Fit test. Prediction by machine learning will be compared with the MDS-UPDRS-III total score and with the 3.14 item (global clinical impression of mobility) of the same scale.
  The patients will be asked to perform all the motor tasks of the MDS-UPDRS-III scale and the finger tapping test (Fit test) with both hands wearing the IMU system.
Objective and subjective mobility | 12 months
  Prediction of mobility by machine learning based on data from IMU wearable sensors; finger tapping test; VAS motor
Sleep and sleepiness | 12 months
  Measured by sleep diary, SSS
Cognition (electronic Stroop test) | 12 months
Emotional state | 12 months
  Measured by Visual Analog Scale(VAS) mood/anxiety
Fatigue | 12 months
  Measured by VAS fatigue
Circadian phase | 12 months
  Continuously for skin body temperature and repeated samples (every 30' for a total of 9 samples, in the evening around the bed time, for salivary DLMO
Sleep homeostasis (SWA) | 12 months
  Calculated based on the EEG recording acquired by means of nocturnal portable polysomnography.

SECONDARY OUTCOMES:
Chronotype | 12 months
  Measured by Horne & Ostberg Morningness/Eveningness Questionnaire (MEQ)
Sleep habits, sleep and wake-related symptoms, sleep quality | 12 months
  Measured by Pittsburgh Sleep Quality Index (PSQI)
PD-specific sleep and wake-associated symptoms | 12 months
  Measured by Parkinson's Disease Sleep Scale (PDSS-2)
Daytime symptoms of bad or insufficient sleep | 12 months
  Measured by Epworth Sleepiness Scale (ESS) [96] and Fatigue Severity Scale (FSS)
Modification of mobility on morning awakening | 12 months
  Measured by Sleep benefit questionnaire
Motor and non-motor symptoms of PD in daily living | 12 months
  Measurded by MDS-UPDRS scale (parts I, II and IV)
Neuropsychological battery useful in idiopathic PD | 12 months
  Measured by Mattis dementia rating scale (MDRS)
Mood | 12 months
  Measured by Beck Depression Inventory (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Luca RATTI, MD, Principal Investigator — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, France

IPD SHARING:
Plan to Share IPD: No